CLINICAL TRIAL: NCT00402519
Title: Interstitial Brachytherapy Alone Versus External Beam Radiation Therapy After Breast Conserving Surgery for Low-risk Invasive Carcinoma and Low-risk Ductal Carcinoma in Situ (DCIS) of the Female Breast
Brief Title: APBI Versus EBRT Therapy After Breast Conserving Surgery for Low-risk Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEC-ESTRO APBI Trial
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: accelerated partial breast irradiation; multicatheter brachytherapy; high dose rate brachytherapy; pulsed dose rate brachytherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- APBI (Experimental): Accelerated Partial Breast Irradiation with multicatheter brachytherapy
  Interventions: Radiation: Accelerated partial breast irradiation
- EBRT (Active Comparator): Standard External Beam Whole Breast Irradiation
  Interventions: Radiation: External beam whole breast irradiation

INTERVENTIONS:
Radiation: Accelerated partial breast irradiation — APBI with PDR and HDR brachytherapy
  Arms: APBI
Radiation: External beam whole breast irradiation — Standard Whole breast irradiation
  Arms: EBRT

SUMMARY:
To assess the role of interstitial brachytherapy alone compared to whole breast irradiation in a defined low-risk group of invasive breast cancer or ductal carcinoma in situ concerning local failure (all ipsilateral local recurrences) to affirm the hypothesis that local control rates in each arm are equivalent.

DETAILED DESCRIPTION:
To assess the role of interstitial brachytherapy alone compared to whole breast irradiation in a defined low-risk group of invasive breast cancer or ductal carcinoma in situ concerning local failure (all ipsilateral local recurrences) to affirm the hypothesis that local control rates in each arm are equivalent.

ELIGIBILITY:
Inclusion Criteria:

* Stage 0, I or II breast cancer.
* Invasive ductal, papillary, mucinous, tubular, medullary or lobular carcinoma.
* Ductal carcinoma in situ (DCIS) alone.
* No lymph invasion (L0) and no hemangiosis (V0).
* Lesions of > 3 cm diameter, histopathologically confirmed.
* pN0/pNmi (a minimum of 6 nodes in specimen, or a negative sentinel node is acceptable); in the case of DCIS alone axillary staging (e.g. sentinel lymph node biopsy) is optional.
* M0.
* Clear resection margins at least 2 mm in any direction; by lobular histology or DCIS histology only the resection margins must be clear at least 5 mm.
* For DCIS only: lesions must be classified as low or intermediate risk group (Van Nuys Prognostic Index <8).
* Unifocal and unicentric DCIS or breast cancer.
* Age >= 40 years.
* Time interval from final definitive breast surgical procedure to the start of external beam therapy or to brachytherapy is less than 12 weeks (84 days). If patients receive chemotherapy the radiotherapy can be started before systemic treatment (within 12 weeks). The radiation therapy can be also given in the interval between the chemotherapy courses. It is also possible to start radiation therapy after chemotherapy is completed according local protocols as soon as possible within 4 weeks after chemotherapy.
* Signed study-specific consent form prior to randomization.

Exclusion Criteria:

* Stage III or IV breast cancer.
* Surgical margins that cannot be microscopically assessed.
* Extensive intraductal component (EIC).
* Paget's disease or pathological skin involvement.
* Synchronous or previous breast cancer.
* Prior malignancy (< 5 years prior to enrollment in study) except non-melanoma skin cancer or cervical carcinoma FIGO 0 and I if patient is continuously disease-free.
* Pregnant or lactating women.
* Collagen vascular disease.
* The presence of congenital diseases with increased radiation sensitivity, for example Ataxia telangiectatica or similar.
* Psychiatric disorders.
* Patient with breast deemed technically unsatisfactory for brachytherapy.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2004-11; Primary Completion 2009-11 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Local control | 5-years, 10 ten-years

SECONDARY OUTCOMES:
Incidence and severity of acute and late side effects | 5-years
Differences in cosmetic results | 5-years
Distant metastases free survival | 5-years
Survival rates (Overall Survival, Disease-free Survival) | 5-years
Contralateral breast cancer rate | 5-years
Quality-of-Life | 5-years

CONTACTS AND LOCATIONS:
Overall Officials: Vratislav Strnad, MD, Study Chair — University Hospital Erlangen, Germany; Csaba Polgár, MD, Study Chair — National Institute of Oncology Budapest, Hungary; Oliver J Ott, MD, Study Director — University Hospital Erlangen, Germany
Locations (11):
- University Hospital AKH Wien, Department of Radiotherapy and Radiobiology, Vienna, Austria
- Germany (6):
  - University Hospital Erlangen, Department of Radiation Oncology, Erlangen
  - University Hospital Kiel, Department of Radiation Oncology, Kiel
  - University Hospital Leipzig, Department of Radiation Oncology, Leipzig
  - University Hospital Lübeck, Department of Radiation Oncology, Lübeck
  - Hospital Barmherzige Brüder, Department of Radiation Oncology, Regensburg
  - University Hospital Rostock, Department of Radiation Oncology, Rostock
- National Institute of Oncology, Department of Radiation Oncology, Budapest, Hungary
- Kierownik Zakladu Brachyterapii, Cetrum Onkologii, Warsaw, Poland
- Spain (2):
  - Catalan Institut of Oncology, Department of Radiation Oncology, Barcelona
  - Valencian Institut of Oncology, Department of Radiation Oncology, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Strnad V, Polgar C, Ott OJ, Hildebrandt G, Kauer-Dorner D, Knauerhase H, Major T, Lyczek J, Guinot JL, Gutierrez Miguelez C, Slampa P, Allgauer M, Lossl K, Polat B, Fietkau R, Schlamann A, Resch A, Kulik A, Arribas L, Niehoff P, Guedea F, Dunst J, Gall C, Uter W; Groupe Europeen de Curietherapie and European Society for Radiotherapy and Oncology. Accelerated partial breast irradiation using sole interstitial multicatheter brachytherapy compared with whole-breast irradiation with boost for early breast cancer: 10-year results of a GEC-ESTRO randomised, phase 3, non-inferiority trial. Lancet Oncol. 2023 Mar;24(3):262-272. doi: 10.1016/S1470-2045(23)00018-9. Epub 2023 Feb 1. PMID 36738756
- [Derived] Schafer R, Strnad V, Polgar C, Uter W, Hildebrandt G, Ott OJ, Kauer-Dorner D, Knauerhase H, Major T, Lyczek J, Guinot JL, Dunst J, Miguelez CG, Slampa P, Allgauer M, Lossl K, Kovacs G, Fischedick AR, Fietkau R, Resch A, Kulik A, Arribas L, Niehoff P, Guedea F, Schlamann A, Gall C, Polat B; Groupe Europeen de Curietherapie of European Society for Radiotherapy and Oncology (GEC-ESTRO). Quality-of-life results for accelerated partial breast irradiation with interstitial brachytherapy versus whole-breast irradiation in early breast cancer after breast-conserving surgery (GEC-ESTRO): 5-year results of a randomised, phase 3 trial. Lancet Oncol. 2018 Jun;19(6):834-844. doi: 10.1016/S1470-2045(18)30195-5. Epub 2018 Apr 22. PMID 29695348
- [Derived] Polgar C, Ott OJ, Hildebrandt G, Kauer-Dorner D, Knauerhase H, Major T, Lyczek J, Guinot JL, Dunst J, Miguelez CG, Slampa P, Allgauer M, Lossl K, Polat B, Kovacs G, Fischedick AR, Fietkau R, Resch A, Kulik A, Arribas L, Niehoff P, Guedea F, Schlamann A, Potter R, Gall C, Uter W, Strnad V; Groupe Europeen de Curietherapie of European Society for Radiotherapy and Oncology (GEC-ESTRO). Late side-effects and cosmetic results of accelerated partial breast irradiation with interstitial brachytherapy versus whole-breast irradiation after breast-conserving surgery for low-risk invasive and in-situ carcinoma of the female breast: 5-year results of a randomised, controlled, phase 3 trial. Lancet Oncol. 2017 Feb;18(2):259-268. doi: 10.1016/S1470-2045(17)30011-6. Epub 2017 Jan 14. PMID 28094198
- [Derived] Ott OJ, Strnad V, Hildebrandt G, Kauer-Dorner D, Knauerhase H, Major T, Lyczek J, Guinot JL, Dunst J, Miguelez CG, Slampa P, Allgauer M, Lossl K, Polat B, Kovacs G, Fischedick AR, Wendt TG, Fietkau R, Kortmann RD, Resch A, Kulik A, Arribas L, Niehoff P, Guedea F, Schlamann A, Potter R, Gall C, Malzer M, Uter W, Polgar C; Groupe Europeen de Curietherapie of European Society for Radiotherapy and Oncology (GEC-ESTRO). GEC-ESTRO multicenter phase 3-trial: Accelerated partial breast irradiation with interstitial multicatheter brachytherapy versus external beam whole breast irradiation: Early toxicity and patient compliance. Radiother Oncol. 2016 Jul;120(1):119-23. doi: 10.1016/j.radonc.2016.06.019. Epub 2016 Jul 12. PMID 27422584
- [Derived] Strnad V, Ott OJ, Hildebrandt G, Kauer-Dorner D, Knauerhase H, Major T, Lyczek J, Guinot JL, Dunst J, Gutierrez Miguelez C, Slampa P, Allgauer M, Lossl K, Polat B, Kovacs G, Fischedick AR, Wendt TG, Fietkau R, Hindemith M, Resch A, Kulik A, Arribas L, Niehoff P, Guedea F, Schlamann A, Potter R, Gall C, Malzer M, Uter W, Polgar C; Groupe Europeen de Curietherapie of European Society for Radiotherapy and Oncology (GEC-ESTRO). 5-year results of accelerated partial breast irradiation using sole interstitial multicatheter brachytherapy versus whole-breast irradiation with boost after breast-conserving surgery for low-risk invasive and in-situ carcinoma of the female breast: a randomised, phase 3, non-inferiority trial. Lancet. 2016 Jan 16;387(10015):229-38. doi: 10.1016/S0140-6736(15)00471-7. Epub 2015 Oct 19. PMID 26494415
- See also: Trial Homepage with a short version of the protocol — http://www.apbi.uni-erlangen.de